CLINICAL TRIAL: NCT00206154
Title: A 6-Month Double-Blind, Double-Dummy, Randomized, Parallel Group, Multicenter Efficacy & Safety Study of SYMBICORT® pMDI 2 x 160/4.5 µg & 80/4.5 µg Bid Compared to Formoterol TBH, Budesonide pMDI (& the Combination) & Placebo in COPD Patients
Brief Title: A Comparison of Symbicort® pMDI 2 x 160/4.5 μg Bid and Symbicort® pMDI 2 x 80/4.5 μg Bid With Formoterol Turbuhaler®, Budesonide pMDI, the Combination of Formoterol Turbuhaler® and Budesonide pMDI, and Placebo in COPD Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D5899C00002; EurodraCT No: 2004-001183-41
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2009-03-27 (Estimated); Status verified 2009-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide

INTERVENTIONS:
Drug: Budesonide/formoterol pMDI
Drug: Budesonide pMDI
Drug: Formoterol Turbuhaler

SUMMARY:
The purpose of this study is to compare a combination asthma drug (Symbicort) with its two components, budesonide and formoterol, taken individually or in combination, and with placebo in the long-term maintenance treatment of patients with chronic obstructive pulmonary disease (COPD)

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of COPD with symptoms for more than 2 years
* Smoking history of 10 or more pack years
* A history of at least one COPD exacerbation requiring a course of oral steroids and/or antibiotics within 1-12 months before first visit.

Exclusion Criteria:

* A history of asthma
* Patients taking oral steroids.
* Any significant disease or disorder that may jeopardize the safety of the patient

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2005-04; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Pre-dose and 1-hour post-dose FEV1 over the 6 months treatment period

SECONDARY OUTCOMES:
Patient-reported outcome variables regarding disease status (incl. PEF), collected via questionnaires and diaries
Health care utilization
Pharmacokinetics (subgroup)
Safety variables, including adverse events, vital signs, ECG, physical examination, hematology, and clinical chemistry.
- all variables assessed over the 6 months treatment period

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Symbicort Medical Science Director, MD, Study Director — AstraZeneca
Locations (212):
- United States (143):
  - Research Site, Birmingham, Alabama
  - Research Site, Jasper, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Glendale, Arizona
  - Research Site, Mesa, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Fort Smith, Arkansas
  - Research Site, Little Rock, Arkansas
  - Research Site, Searcy, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Fullerton, California
  - Research Site, Irvine, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Mission Viejo, California
  - Research Site, Orange, California
  - Research Site, Rancho Cordova, California
  - Research Site, Riverside, California
  - Research Site, San Diego, California
  - Research Site, San Jose, California
  - Research Site, Sepulveda, California
  - Research Site, Signal Hill, California
  - Research Site, Stockton, California
  - Research Site, Torrance, California
  - Research Site, Walnut Creek, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Wheat Ridge, Colorado
  - Research Site, Bristol, Connecticut
  - Research Site, Waterbury, Connecticut
  - Research Site, Bay Pines, Florida
  - Research Site, Brandon, Florida
  - Research Site, Clearwater, Florida
  - Research Site, DeLand, Florida
  - Research Site, Largo, Florida
  - Research Site, Miami Beach, Florida
  - Research Site, Naples, Florida
  - Research Site, Ocala, Florida
  - Research Site, Ormond Beach, Florida
  - Research Site, Panama City, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Port Orange, Florida
  - Research Site, Sarasota, Florida
  - Research Site, Blairsville, Georgia
  - Research Site, Blue Ridge, Georgia
  - Research Site, Marietta, Georgia
  - Research Site, Rome, Georgia
  - Research Site, Coeur d'Alene, Idaho
  - Research Site, Bloomington, Illinois
  - Research Site, Chicago, Illinois
  - Research Site, Hines, Illinois
  - Research Site, Normal, Illinois
  - Research Site, North Chicago, Illinois
  - Research Site, O'Fallon, Illinois
  - Research Site, Evansville, Indiana
  - Research Site, South Bend, Indiana
  - Research Site, Iowa City, Iowa
  - Research Site, Waterloo, Iowa
  - Research Site, Mission, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Lebanon, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Madisonville, Kentucky
  - Research Site, Paducah, Kentucky
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Lafayette, Louisiana
  - Research Site, Marrero, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Sunset, Louisiana
  - Research Site, Auburn, Maine
  - Research Site, Bangor, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Taunton, Massachusetts
  - Research Site, Minneapolis, Minnesota
  - Research Site, Plymouth, Minnesota
  - Research Site, Saint Paul, Minnesota
  - Research Site, Chesterfield, Missouri
  - Research Site, Saint Charles, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Butte, Montana
  - Research Site, Missoula, Montana
  - Research Site, Omaha, Nebraska
  - Research Site, Papillion, Nebraska
  - Research Site, Scottsbluff, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Pahrump, Nevada
  - Research Site, Reno, Nevada
  - Research Site, Cherry Hill, New Jersey
  - Research Site, Skillman, New Jersey
  - Research Site, Springfield, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Bay Shore, New York
  - Research Site, Buffalo, New York
  - Research Site, Larchmont, New York
  - Research Site, Mineola, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Bismarck, North Dakota
  - Research Site, Akron, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Mogadore, Ohio
  - Research Site, Sylvania, Ohio
  - Research Site, Zanesville, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Eugene, Oregon
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Easton, Pennsylvania
  - Research Site, Erie, Pennsylvania
  - Research Site, Hershey, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Ridley Park, Pennsylvania
  - Research Site, Swarthmore, Pennsylvania
  - Research Site, West Chester, Pennsylvania
  - Research Site, East Providence, Rhode Island
  - Research Site, Charleston, South Carolina
  - Research Site, Simpsonville, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Austin, Texas
  - Research Site, Barker, Texas
  - Research Site, Dallas, Texas
  - Research Site, El Paso, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, Killeen, Texas
  - Research Site, New Braunfels, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Abingdon, Virginia
  - Research Site, Charlottesville, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Salem, Virginia
  - Research Site, Virginia Beach, Virginia
  - Research Site, Bellingham, Washington
  - Research Site, Seattle, Washington
  - Research Site, Spokane, Washington
  - Research Site, Tacoma, Washington
  - Research Site, La Crosse, Wisconsin
- Czechia (19):
  - Research Site, Prague, CZ
  - Research Site, Ústí nad Labem, CZ
  - Research Site, Beroun
  - Research Site, Cvikov
  - Research Site, Jarom¿¿
  - Research Site, Karlovy Vary
  - Research Site, Kladno
  - Research Site, Kutná Hora
  - Research Site, Liberec
  - Research Site, Lovosice
  - Research Site, Neratovice
  - Research Site, Olomouc
  - Research Site, Ostrava
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Rokycany
  - Research Site, Strakonice
  - Research Site, Ústí nad Labem
  - Research Site, Znojmo
- Netherlands (12):
  - Research Site, Almelo
  - Research Site, Arnhem
  - Research Site, Breda
  - Research Site, Eindhoven
  - Research Site, Groningen
  - Research Site, Harderwijk
  - Research Site, Heerlen
  - Research Site, Nieuwegein
  - Research Site, Terneuzen
  - Research Site, The Hague
  - Research Site, Tilburg
  - Research Site, Utrecht
- Poland (28):
  - Research Site, Bia¿ystok
  - Research Site, Bydgoszcz
  - Research Site, Bystra ¿l¿ska
  - Research Site, Chrzanów
  - Research Site, Ch¿ciny
  - Research Site, Cz¿stochowa
  - Research Site, Gidle
  - Research Site, Gorzów Wlkp
  - Research Site, I¿awa
  - Research Site, Karpacz
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Ostrów Wielkopolski
  - Research Site, Otowck
  - Research Site, Późna
  - Research Site, Proszowice
  - Research Site, Radom
  - Research Site, Siedlce
  - Research Site, Sopot
  - Research Site, Szczecin
  - Research Site, Tarnów
  - Research Site, Turek
  - Research Site, Warsaw
  - Research Site, Wo¿omin
  - Research Site, Zabrze
  - Research Site, Zawadzkie
  - Research Site, ¿om¿a
  - Research Site, ¿ód¿
- South Africa (10):
  - Research Site, Parow, Cape Province
  - Research Site, Lenasia, Gauteng
  - Research Site, Pretoria, Gauteng
  - Research Site, Witbank, Gauteng
  - Research Site, Cape Town, Western Cape
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, eMkhomazi
  - Research Site, Lyttelton Manor
  - Research Site, Port Elizabeth

REFERENCES:
- [Derived] Bafadhel M, Peterson S, De Blas MA, Calverley PM, Rennard SI, Richter K, Fageras M. Predictors of exacerbation risk and response to budesonide in patients with chronic obstructive pulmonary disease: a post-hoc analysis of three randomised trials. Lancet Respir Med. 2018 Feb;6(2):117-126. doi: 10.1016/S2213-2600(18)30006-7. Epub 2018 Jan 10. PMID 29331313
- [Derived] Make BJ, Eriksson G, Calverley PM, Jenkins CR, Postma DS, Peterson S, Ostlund O, Anzueto A. A score to predict short-term risk of COPD exacerbations (SCOPEX). Int J Chron Obstruct Pulmon Dis. 2015 Jan 27;10:201-9. doi: 10.2147/COPD.S69589. eCollection 2015. PMID 25670896
- [Derived] Bleecker ER, Meyers DA, Bailey WC, Sims AM, Bujac SR, Goldman M, Martin UJ. ADRB2 polymorphisms and budesonide/formoterol responses in COPD. Chest. 2012 Aug;142(2):320-328. doi: 10.1378/chest.11-1655. PMID 22383665